CLINICAL TRIAL: NCT07171827
Title: A Prospective Study Comparing Anti CD30 (Brentuximab Vedotin) With AVD Versus ABVD Chemotherapy Protocol Frontline Therapy in Patients With Advanced Classical Hodgkin Lymphoma
Brief Title: Anti-CD30 (Brentuximab Vedotin) With AVD Versus ABVD Chemotherapy Protocol Frontline Therapy in Patients With Advanced Classical Hodgkin Lymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Marwa Nazih Abdel Gawad, Assistant Lecturer of Clinical Oncology, Faculty of Medicine, Helwan University, Egypt., Helwan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 40-2023
Record Dates: First submitted 2025-09-06; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Anti-CD30; Brentuximab; Doxorubicin; Vinblastine; Dacarbazine; Frontline; Advanced Classical Hodgkin Lymphoma
MeSH Terms: interventions — Brentuximab Vedotin; Doxorubicin; Vinblastine; Dacarbazine; Bleomycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BV+AVD group (Experimental): Patients received Brentuximab Vedotin (BV)+ Doxorubicin, Vinblastine, and Dacarbazine (AVD) drug regimen by intravenous infusion on Days 1 and 15 of each 28-day cycle.
  Interventions: Drug: Brentuximab Vedotin + Doxorubicin, Vinblastine, and Dacarbazine
- ABVD group (Experimental): Patients received Doxorubicin, Bleomycin, Vinblastine, and Dacarbazine (ABVD) drug regimen by intravenous infusion on Days 1 and 15 of each 28-day cycle.
  Interventions: Drug: Doxorubicin, Bleomycin, Vinblastine, and Dacarbazine

INTERVENTIONS:
Drug: Brentuximab Vedotin + Doxorubicin, Vinblastine, and Dacarbazine — Patients received Brentuximab Vedotin (BV)+ Doxorubicin, Vinblastine, and Dacarbazine (AVD) drug regimen by intravenous infusion on Days 1 and 15 of each 28-day cycle.
  Arms: BV+AVD group
Drug: Doxorubicin, Bleomycin, Vinblastine, and Dacarbazine — Patients received Doxorubicin, Bleomycin, Vinblastine, and Dacarbazine (ABVD) drug regimen by intravenous infusion on Days 1 and 15 of each 28-day cycle.
  Arms: ABVD group

SUMMARY:
This study will be held in the clinical oncology department, Helwan University, and Police Hospital, aiming to compare the efficacy and safety of anti-CD30 (BV) + Doxorubicin, Vinblastine, and Dacarbazine (AVD) versus the standard of care Doxorubicin, Bleomycin, Vinblastine, and Dacarbazine (ABVD) as frontline therapy in patients with advanced classical Hodgkin lymphoma.

DETAILED DESCRIPTION:
Hodgkin lymphoma (HL) is a malignancy that typically originates from germinal center B-lymphocytes. It is subdivided into classical type, which represents 95% of histopathology of HL cases (with four histological subtypes, namely, nodular sclerosis, mixed-cellularity, lymphocyte-rich, and lymphocyte-depleted), and nodular lymphocyte-predominant HL.

For patients with newly diagnosed Ann Arbor stage III/IV (advanced stage) HL, 70% are expected to be cured after treatment with Doxorubicin, Bleomycin, Vinblastine, and Dacarbazine (ABVD), which has been the preferred standard of care in the United States for many years.

The Risk-adapted therapy for advanced-stage Hodgkin lymphoma (RATHL) study assessed de-escalation to Doxorubicin, Vinblastine, and Dacarbazine (AVD) in patients with stage IIB, III, or IV HL (Deauville 1-3) and found that positron emission tomography (PET)-adapted de-escalation to AVD failed to demonstrate noninferiority compared with ABVD.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18- 70 Years.
* Histopathology: confirmed classical Hodgkin Lymphoma according to the current World Health Organization (WHO) classification. CD30 positive by immunohistochemistry.
* Stage III or IV Hodgkin lymphoma (HL) by the Ann Arbor classification system.
* Treatment-naïve.
* Laboratory:

  * complete blood count: absolute neutrophil counts (≥1500 per cubic millimeter), platelet counts (≥75,000 per cubic millimeter), and hemoglobin levels (≥8 g per deciliter) (except for patients with involvement of the marrow).
  * liver function test: total bilirubin level <1.5 times the upper limit of normal and alanine aminotransferase or aspartate aminotransferase levels <3 times the upper limit of normal.
  * kidney function test: serum creatinine level, <2.0 mg per deciliter or creatinine clearance or calculated creatinine clearance, >40 ml per minute.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.

Exclusion Criteria:

* Histopathology: Nodular lymphocyte predominant Hodgkin lymphoma and non-Hodgkin lymphoma.
* Cerebral/meningeal disease.
* Prior treatment with chemotherapy, radiotherapy, or any immunotherapy within 12 weeks of first study drug dose.
* Known human immunodeficiency virus (HIV) positive, known hepatitis B surface antigen-positive, or known active hepatitis C infection.
* Known organ failure.
* Cardiac: left ventricular ejection fraction < 50%, myocardial infarction within 2 years of randomization or current uncontrolled cardiovascular conditions, including arrhythmias, congestive heart failure, angina, evidence of acute ischemia, or active conduction system abnormalities.
* Female patients who are breastfeeding or having a positive serum pregnancy test during the randomization period or on day 1 before starting treatment.
* Neurotoxicity, including symptomatic neurologic disease, comprising normal daily activities, any sensory or motor peripheral neuropathy.
* Pulmonary diffusion capacity >25 % lower than predicted value as retrieved by pulmonary function test for each patient before randomization.
* Known hypersensitivity to recombinant proteins, murine proteins, or any component of the included drugs formulation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 2 years post-procedure
  Progression-free Survival was recorded.

SECONDARY OUTCOMES:
Overall response rate | 30 days after the end of treatment
  Overall Response Rate (ORR) is the percentage of participants who achieved complete remission (CR) or partial remission (PR) at the end of treatment with randomized regimen.
Overall survival | 2 years post-procedure
  Overall survival was recorded.
Incidence of adverse events | 30 days after the end of frontline therapy
  Incidence of adverse events such as toxicity, incidence, severity and type starting after administration of the first dose till 30 days after end of frontline therapy were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Helwan University, Helwan, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.